CLINICAL TRIAL: NCT01315353
Title: A Randomized Trial To Compare An HPV Test-And-Treat Strategy To A Cytology-Based Strategy For Prevention Of CIN 2+ In HIV-Infected Women
Brief Title: HPV Test-and-Treat-Strategy Versus Cytology-based Strategy for Prevention of CIN2+ in HIV-Infected Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5282; 1U01AI068636 (NIH)
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: Immediate cryotherapy (HPV test-and-treat) (Experimental): Participants in Arm A (HPV test-and-treat) had cervical cryotherapy at entry. Post entry, participants in Arm A were seen at regular intervals for the collection of cervical specimens, cytology, and as needed, cervical colposcopy, directed biopsies, and LEEP.
  Interventions: Procedure: Cervical Cryotherapy; Procedure: Loop Electrosurgical Excision Procedure (LEEP)
- Arm B: cytology-based strategy (Experimental): Participants in Arm B followed a cytology-based management plan involving three steps- cytology, colposcopy with directed biopsies, and LEEP (as needed).
  Interventions: Procedure: Loop Electrosurgical Excision Procedure (LEEP)
- Arm C : Ineligible for randomization to Arm A or B (Experimental): Participants were eligible for Arm C under the conditions noted in the inclusion criteria. Participants in Arm C had colposcopy and directed biopsies at entry. If CIN2+ was found by biopsy, then LEEP was performed and a follow-up visit 26 weeks after these procedures was scheduled for the collection of cervical specimens, cytology, and as needed, cervical colposcopy, directed biopsies, and LEEP. After the week 26 visit, Arm C participants went off study.
  Interventions: Procedure: Loop Electrosurgical Excision Procedure (LEEP)

INTERVENTIONS:
Procedure: Cervical Cryotherapy — Participants had cervical cryotherapy within 7 days after study entry. The cryotherapy consists of two 3-minute freezes separated by 5 minutes of thawing.
  Arms: Arm A: Immediate cryotherapy (HPV test-and-treat)
Procedure: Loop Electrosurgical Excision Procedure (LEEP) — Loop Electrosurgical Excision Procedure (LEEP): Participants found to have CIN2+ by biopsy had LEEP, an electro-surgical procedure used to treat high-grade cervical dysplasia.

SUMMARY:
Women sometimes develop cancer in an area called the cervix, which is the opening to the uterus, or womb. Women who have HIV are more likely to get this kind of cancer than women who do not have HIV. Nearly all of these cancers are caused by another virus, called human papilloma virus (or HPV). Other times, the cause of this cancer is not known.

The investigators are looking for a better way to prevent cervical cancer. This study is comparing two different methods to prevent cancer of the cervix in women who have HIV. This study will also see if these methods are safe and tolerable in women who have HIV.

DETAILED DESCRIPTION:
The study had two components:

1. a randomized open-label comparison between immediate cryotherapy (test-and-treat strategy; Arm A) and cytology-based strategy (Arm B) in participants detected with high-risk HPV (hr-HPV), and
2. a brief cohort follow-up for participants for whom cryotherapy was inappropriate (Arm C).

The study's primary objective was to evaluate the effectiveness of immediate cryotherapy (Arm A) compared to the cytology-based strategy (Arm B).

The total target sample size was up to 450 (280 for Arms A and B, approximately 170 for Arm C). Randomization to Arms A and B was stratified by use of antiretroviral therapy (ART) at screening (taking any ART or not taking any ART) with institutional balancing.

All study participants were screened with the Abbott RealTime hr-HPV test (aHPV) to detect hr-HPV infection.

At screening, the examiner also performed a visual inspection and colposcopy without biopsies to determine whether the candidate's cervix was suitable for cryotherapy (see inclusion criteria for definition).

Participants with cervical lesions inappropriate for cryotherapy were not eligible for randomization (to Arms A or B) but were eligible to register to Arm C. Participants without hr-HPV (by aHPV) were also eligible to register to Arm C if lesions were seen on the screening colposcopy or if the screening cytology showed high-grade squamous intraepithelial lesions (HSIL). Arm C provided a larger number of participants for assessments of HPV genotypes found in CIN2+ (cervical intraepithelial neoplasia grade 2, 3, or invasive cancer) biopsy specimens and of the effect of LEEP on prevalent hr-HPV infections. In addition, Arm C provided important data for implementation of the HPV test-and-treat strategy including the role of HPV testing in the management of women with extensive cervical lesions inappropriate for cervical cryotherapy, hr-HPV negative women with cervical lesions or HSIL cytology.

Participants in Arm A undergo one or two cervical biopsies followed by immediate cervical cryotherapy at entry. Up to two visible lesions were biopsied. If no lesions were seen, then one normal-appearing area of the cervix was biopsied. Participants in Arm A received the results of the biopsy, but participants received cryotherapy treatment regardless of the results.

Participants in Arm B followed a cytology-based management plan involving three steps - cytology, colposcopy with directed biopsies, and loop electrosurgical excision procedure (LEEP), as needed.

Participants in Arms A and B were seen at weeks 26, 52, 78, 104 and 130 post entry for evaluation using aHPV, HPV DNA PCR, cervical cytology, and cervical colposcopy and directed biopsies for a total follow-up length of 130 weeks. Biopsies were expected for participants with abnormal cytology and with visible cervical lesions on colposcopy.

Participants in Arm C undergo colposcopy and directed biopsies. If CIN2+ was detected by biopsy, then LEEP was performed and a follow-up visit 26 weeks after these procedures was scheduled for evaluation using aHPV, HPV DNA PCR, Xpert HPV, cervical cytology, and cervical colposcopy and directed biopsies. After the week 26 visit, Arm C participants went off study.

All participants who had cryotherapy or LEEP were seen 4 weeks post-procedure to evaluate potential adverse events (AEs) from the procedure.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection.
* Certain laboratory values obtained within 45 days prior to study entry (more information can be found in the protocol).
* For candidates suitable for cervical cryotherapy, hr-HPV detected by aHPV within 45 days prior to study entry.
* For women without hr-HPV detected by the aHPV assay, presence of lesions on visual inspection or HSIL cervical cytology. These participants are not eligible for randomization to Arms A or B and were followed in Arm C.
* Suitable candidate for cervical cryotherapy (as defined in the protocol): No visible cervical lesions, OR (a) any visible lesions were located entirely on the ectocervix and were no more than 2 to 3 mm. into the endocervical canal, AND (b) visible lesions covered less than 75% of the cervix, AND (c) all visible lesions were deemed appropriate for cryotherapy by the treating local health care provider.

NOTE: Participants with cervical lesions inappropriate for cryotherapy are not eligible for randomization to Arms A or B and were followed in Arm C.

* For participants of reproductive potential, negative pregnancy test within 48 hours prior to study entry.
* Must agree not to participate in a conception process (e.g. active attempt to get pregnant or in vitro fertilization), or use at least one reliable contraceptive if participating in sexual activity, from time of study entry until 12 weeks after study entry.
* If recently gave birth, must be at least 12 weeks postpartum.
* Ability and willingness of participant or legal guardian/representative to provide written informed consent.

Exclusion Criteria:

* Current or prior history of cervical, vaginal, or vulvar cancer.
* Prior cervical cryotherapy, LEEP, cervical conization, or total or partial hysterectomy.
* Cervical, vaginal, or vulvar lesions that are suspicious on clinical exam for cancer.
* Visual evidence of bacterial STIs (sexually transmitted infections) or suspicion of pelvic inflammatory disease.
* Prior vaccination with an HPV vaccine.
* Hemophilia.
* Currently on anticoagulation therapy other than acetylsalicylic acid.
* Serious illness requiring systemic treatment and/or hospitalization within 21 days prior to study entry.
* Active drug or alcohol use or dependence or any other condition that, in the opinion of the site investigator, would interfere with the participant's ability to adhere to study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2012-04-04 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Wilkin, MD, MPH, Study Chair — Cornell Clinical Research Site
Locations (13):
- Botswana (2):
  - Gaborone Prevention/Treatment Trials CRS (12701), Gaborone
  - Molepolole Prevention/Treatment Trials CRS (12702), Molepolole
- Les Centres GHESKIO CRS (30022), Port-au-Prince, Haiti
- India (2):
  - BJ Medical College CRS (31441), Pune, Maharashtra
  - National AIDS Research Institute Pune CRS (11601), Pune, Maharashtra
- Malawi (2):
  - College of Med. JHU CRS (30301), Blantyre
  - University of North Carolina Lilongwe CRS (12001), Lilongwe
- Peru (2):
  - Investigaciones Medicas en Salud (INMENSA) (11302), San Isidro, Lima region
  - Asociacion Civil Impacta Salud y Educacion - Miraf CRS (11301), Lima
- South Africa (3):
  - Durban Adult HIV CRS (11201), Durban
  - Soweto ACTG CRS (12301), Johannesburg
  - Univ. of Witwatersrand CRS (11101), Johannesburg
- UZ-Parirenyatwa CRS (30313), Harare, Zimbabwe

REFERENCES:
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004; Clarification, August 2009. — https://rsc.tech-res.com/docs/default-source/safety/table_for_grading_severity_of_adult_pediatric_adverse_events.pdf?sfvrsn=6
- See also: Addendum 1 Female Genital Grading Table for Use in Microbicide Studies — https://rsc.tech-res.com/docs/default-source/safety/addendum_1_female_genital_grading_table_v1_nov_2007.pdf?sfvrsn=8
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.tech-res.com/docs/default-source/safety/manual_for_expedited_reporting_aes_to_daids_v2.pdf?sfvrsn=10

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from April 2012 to June 2014 from 7 different countries.
Groups:
- Arm A: Immediate Cryotherapy (HPV Test-and-treat): Participants in Arm A (HPV test-and-treat) had cervical cryotherapy at entry. Post entry, participants in Arm A were seen at regular intervals for the collection of cervical specimens, cytology, and as needed, cervical colposcopy, directed biopsies, and LEEP.
  Cervical Cryotherapy: Participants had cervical cryotherapy within 7 days after study entry. The cryotherapy consists of two 3-minute freezes separated by 5 minutes of thawing.
  Loop Electrosurgical Excision Procedure (LEEP): Participants found to have CIN2+ by biopsy post-entry had LEEP, an electro-surgical procedure used to treat high-grade cervical dysplasia.
- Arm B: Cytology-based Strategy: Participants in Arm B followed a cytology-based management plan involving three steps- cytology, colposcopy with directed biopsies, and LEEP (as needed).
  Loop Electrosurgical Excision Procedure (LEEP): Participants found to have CIN2+ by biopsy at any point during the study had LEEP, an electro-surgical procedure used to treat high-grade cervical dysplasia.
- Arm C : Ineligible for Randomization to Arm A or B: Participants were eligible for Arm C under the conditions noted in the inclusion criteria. Participants in Arm C had colposcopy and directed biopsies at entry. If CIN2+ is found by biopsy, then LEEP was performed and a follow-up visit 26 weeks after these procedures was scheduled for the collection of cervical specimens, cytology, and as needed, cervical colposcopy, directed biopsies, and LEEP. After the week 26 visit, Arm C participants went off study.
  Loop Electrosurgical Excision Procedure (LEEP): Participants found to have CIN2+ by biopsy at any point during the study had LEEP, an electro-surgical procedure used to treat high-grade cervical dysplasia.
Period: Overall Study
Arm/Group | Arm A: Immediate Cryotherapy (HPV Test-and-treat) | Arm B: Cytology-based Strategy | Arm C : Ineligible for Randomization to Arm A or B
Started | 145 | 143 | 179
Completed | 116 | 120 | 166
Not Completed | 29 | 23 | 13
Not completed — Death | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 6 | 1
Not completed — Lost to Follow-up | 13 | 6 | 6
Not completed — Unwilling to adhere to requirements | 5 | 5 | 4
Not completed — Site closing | 7 | 4 | 0
Not completed — Taken off study by site in error | 0 | 1 | 0
Not completed — Inadvertent randomization/assignment | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat: All eligible participants were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Immediate Cryotherapy (HPV Test-and-treat) | Arm B: Cytology-based Strategy | Arm C : Ineligible for Randomization to Arm A or B | Total
Number analyzed (Participants) | 145 | 143 | 177 | 465
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 145 | 143 | 175 | 463
  >=65 years | 0 | 0 | 2 | 2
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [32 to 42] | 34 [29 to 39] | 36 [32 to 42] | 36 [31 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 143 | 177 | 465
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Non-Hispanic | 106 | 107 | 156 | 369
  Hispanic (Regardless of Race) | 11 | 9 | 6 | 26
  Asian, Pacific Islander | 28 | 27 | 15 | 70
Region of Enrollment [Count of Participants; unit: Participants]
  Haiti | 3 | 3 | 16 | 22
  Malawi | 35 | 37 | 23 | 95
  Botswana | 8 | 7 | 45 | 60
  South Africa | 40 | 41 | 55 | 136
  Zimbabwe | 20 | 19 | 17 | 56
  Peru | 11 | 9 | 6 | 26
  India | 28 | 27 | 15 | 70
CD4+ T-cell Count [Median (Inter-Quartile Range); unit: cells/mm^3] — CD4+ T-cell count at entry. Population: Includes participants with non-missing entry CD4+ T-cell counts.
  cells/mm^3
    number analyzed (Participants) | 108 | 106 | 146 | 360
    (all) | 529 [386 to 687] | 479 [330 to 649] | 568 [391 to 728] | 521 [381 to 699]
Nadir CD4+ T-Cell Count [Count of Participants; unit: Participants] — Nadir CD4+ T-cell count at screening. Population: Included participants with non-missing nadir CD4+ T-cell count.
  Participants
    number analyzed (Participants) | 134 | 135 | 167 | 436
    <=50 cells/mm^3 | 16 | 15 | 13 | 44
    51-100 cells/mm^3 | 12 | 19 | 17 | 48
    101-200 cells/mm^3 | 33 | 34 | 34 | 101
    201-500 cells/mm^3 | 61 | 57 | 70 | 188
    >500 cells/mm^3 | 12 | 10 | 33 | 55
HIV-1 RNA [Count of Participants; unit: Participants] — Entry HIV-1 RNA value categorized as below the assay's corresponding lower limit of quantification (<LLQ) or otherwise (>=LLQ).
  Participants
    <LLQ | 93 | 85 | 116 | 294
    >=LLQ | 52 | 58 | 61 | 171
Antiretroviral Therapy (ART) Use [Count of Participants; unit: Participants] — Participants status of ART use at screening.
  Participants
    Not taking any ART | 25 | 22 | 35 | 82
    Taking any ART | 120 | 121 | 142 | 383

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Rate of Cervical Intraepithelial Neoplasia (CIN2+) (CIN2, CIN3 or Invasive Cancer) by Week 130
Description: The Kaplan-Meier estimate of the cumulative rate of CIN2+ (CIN2, CIN3 or invasive cancer) by week 130.
  Time to CIN2+ was computed as the number of weeks between randomization and the week 26 to week 130 biopsy week when CIN2+ was first detected. For those who did not develop CIN2+, event time was censored at the latest among the following: time of last biopsy or last colposcopy or last pap smear. CIN2+ diagnosis by biopsy was determined by local review at a DAIDS-assessed laboratory.
Time Frame: Weeks 26, 52, 78, 104 and 130 post randomization
Population: Intent to treat: All eligible participants were included in the analysis: participants were analyzed per original assigned randomized treatment. Analysis was limited to the two randomized study arms (Arms A and B).
Measure: Number (95% Confidence Interval); unit: Events per 100 persons
Arm/Group | Arm A: Immediate Cryotherapy (HPV Test-and-treat) | Arm B: Cytology-based Strategy
Number analyzed (Participants) | 145 | 143
Events per 100 persons | 24.9 [16.9 to 32.9] | 26.5 [18.3 to 34.7]
Statistical Analysis 1: Comparison: Arm A: Immediate Cryotherapy (HPV Test-and-treat) vs Arm B: Cytology-based Strategy; Treatment comparison was made using the difference (arm B - arm A) in the stratified Kaplan-Meier estimate for the week 130 cumulative rate of CIN2+ with 95% one-sided confidence interval; Test type: Superiority — Confidence interval estimation was stratified by ART use at screening using Greenwood's variance with the inverse of this variance used for the stratum weights; Cumulative rate difference = 1.7, 95% CI 1-sided [lower limit -7.9] — The lower bound of the (lower) one-sided 95% confidence interval was provided

2. Secondary Outcome: Time to CIN2+ Diagnosis by Biopsy, as Determined by Local Review at a DAIDS-assessed Laboratory.
Description: Time to CIN2+ was computed as the number of weeks between randomization and the week 26 to week 130 biopsy week when CIN2+ was first detected. For those who did not develop CIN2+, event time was censored at the latest among the following: time of last biopsy or last colposcopy or last pap smear. The 10th percentile of the time to CIN2+ (the number of weeks at which 10% of participants had had CIN2+ diagnosis) is presented in the data table below.
Time Frame: Weeks 26, 52, 78, 104 and 130 post randomization
Population: Intent to treat: All eligible participants were included in the analysis. Analysis was limited to the two randomized study arms (Arms A and B).
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Arm A: Immediate Cryotherapy (HPV Test-and-treat) | Arm B: Cytology-based Strategy
Number analyzed (Participants) | 145 | 143
weeks | 31 [28 to 66] | 30 [27 to 87]
Statistical Analysis 1: Comparison: Arm A: Immediate Cryotherapy (HPV Test-and-treat) vs Arm B: Cytology-based Strategy; Null Hypothesis: There is no difference between Arm A and Arm B with respect to time to CIN2+; Test type: Other; p = 0.94, Log Rank — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance used for the two-sided test was 0.05; Log-rank test was stratified by ART use at screening

3. Secondary Outcome: Cumulative Rate of CIN3+ (CIN3 or Invasive Cancer) by Week 130.
Description: The Kaplan-Meier estimate of the cumulative rate of CIN3+ (CIN3 or invasive cancer) by week 130.
  Time to CIN3+ was computed as the number of weeks between randomization and the week 26 to week 130 biopsy week when CIN3+ was first detected. For those who did not develop CIN3+, event time was censored at the latest among the following: time of last biopsy or last colposcopy or last pap smear. CIN3+ diagnosis by biopsy was determined by local review at a DAIDS-assessed laboratory.
Time Frame: Weeks 26, 52, 78, 104 and 130 post randomization
Population: Intent-to-treat: All eligible participants were included in the analysis: participants were analyzed per original assigned randomized treatment. Analysis was limited to the two randomized study arms (Arms A and B).
Measure: Number (95% Confidence Interval); unit: Cumulative rate of events/100 persons
Arm/Group | Arm A: Immediate Cryotherapy (HPV Test-and-treat) | Arm B: Cytology-based Strategy
Number analyzed (Participants) | 145 | 143
Cumulative rate of events/100 persons | 12.7 [6.8 to 18.6] | 17.1 [10.0 to 24.3]
Statistical Analysis 1: Comparison: Arm A: Immediate Cryotherapy (HPV Test-and-treat) vs Arm B: Cytology-based Strategy; Treatment comparison was made using the difference (arm B - arm A) in the stratified Kaplan-Meier estimate for the week 130 cumulative rate of CIN3+ with 95% two-sided confidence interval; Test type: Other; Cumulative rate difference = 4.4, 95% CI 2-sided [-4.8 to 13.6] — Confidence interval estimation was stratified by ART use at screening using Greenwood's variance with the inverse of this variance used for the stratum weights

4. Secondary Outcome: Number of Participants Who Discontinued Study Early.
Description: The number of participants who did not complete the study.
Time Frame: 0 to 130 weeks post randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Immediate Cryotherapy (HPV Test-and-treat) | Arm B: Cytology-based Strategy
Number analyzed (Participants) | 145 | 143
Participants | 29 | 23
Statistical Analysis 1: Comparison: Arm A: Immediate Cryotherapy (HPV Test-and-treat) vs Arm B: Cytology-based Strategy; Null hypothesis: There is no difference between Arm A and Arm B with respect to rate of premature study discontinuation; Test type: Other; p = 0.445, Fisher Exact — [p-value comment as in outcome 2, analysis 1]

5. Secondary Outcome: Number of Participants With Abnormal Cytology Results at Study Visits.
Description: Number of participants with abnormal (ASCUS: atypical squamous cells; undetermined significance, ASC-H: atypical squamous cells; favor high-grade squamous intra-epithelial lesion, LSIL: low-grade squamous intraepithelial lesion/mild dysplasia/HPV, HSIL: high-grade squamous intraepithelial lesion/moderate or severe dysplasia/carcinoma in situ/features of invasion; squamous cell carcinoma) cytology results.
Time Frame: Weeks 26, 52, 78, 104 and 130 post randomization
Population: Included participants with available cytology results.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Immediate Cryotherapy (HPV Test-and-treat) | Arm B: Cytology-based Strategy
Number analyzed (Participants) | 145 | 143
Participants
  Week 26: With Abnormal Cytology: number analyzed (Participants) | 123 | 116
  Week 26: With Abnormal Cytology | 80 | 75
  Week 52: With Abnormal Cytology: number analyzed (Participants) | 118 | 119
  Week 52: With Abnormal Cytology | 80 | 72
  Week 78: With Abnormal Cytology: number analyzed (Participants) | 107 | 105
  Week 78: With Abnormal Cytology | 63 | 64
  Week 104: With Abnormal Cytology: number analyzed (Participants) | 97 | 95
  Week 104: With Abnormal Cytology | 57 | 62
  Week 130: With Abnormal Cytology: number analyzed (Participants) | 76 | 93
  Week 130: With Abnormal Cytology | 33 | 46
Statistical Analysis 1: Comparison: Arm A: Immediate Cryotherapy (HPV Test-and-treat) vs Arm B: Cytology-based Strategy; Null Hypothesis: There is no difference between Arm A and Arm B with respect to the proportion of participants with abnormal cervical cytology results at week 26; Test type: Other; p = 1.000, Fisher Exact — P-value for the week 26 comparison. The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance used for the two-sided test was 0.05
Statistical Analysis 2: Comparison: Arm A: Immediate Cryotherapy (HPV Test-and-treat) vs Arm B: Cytology-based Strategy; Null Hypothesis: There is no difference between the Arm A and Arm B with respect to the proportion of participants with abnormal cervical cytology results at week 52; Test type: Other; p = 0.279, Fisher Exact — P-value for the week 52 comparison. The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance used for the two-sided test was 0.05
Statistical Analysis 3: Comparison: Arm A: Immediate Cryotherapy (HPV Test-and-treat) vs Arm B: Cytology-based Strategy; Null Hypothesis: There is no difference between Arm A and Arm B with respect to the proportion of participants with abnormal cervical cytology results at week 78; Test type: Other; p = 0.781, Fisher Exact — P-value for the week 78 comparison. The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance used for the two-sided test was 0.05
Statistical Analysis 4: Comparison: Arm A: Immediate Cryotherapy (HPV Test-and-treat) vs Arm B: Cytology-based Strategy; Null Hypothesis: There is no difference between Arm A and Arm B with respect to the proportion of participants with abnormal cervical cytology results at week 104; Test type: Other; p = 0.375, Fisher Exact — P-value for the week 104 comparison. The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance used for the two-sided test was 0.05
Statistical Analysis 5: Comparison: Arm A: Immediate Cryotherapy (HPV Test-and-treat) vs Arm B: Cytology-based Strategy; Null Hypothesis: There is no difference between Arm A and Arm B with respect to the proportion of participants with abnormal cervical cytology results at week 130; Test type: Other; p = 0.444, Fisher Exact — P-value for the week 130 comparison. The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance used for the two-sided test was 0.05

6. Secondary Outcome: Number of Participants With High Risk (hr)-HPV by the Abbott Real Time High-risk HPV Assay (aHPV) at Study Visits.
Description: Number of participants with hr-HPV (HPV 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, 68) as detected by the Abbott Real Time high-risk HPV assay. Specimens for weeks 52, 78, 104 and 130 were not tested due to insufficient funding.
Time Frame: Weeks 26, 52, 78, 104 and 130 post randomization
Population: Includes participants with results for Abbott Real Time high-risk HPV assay
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Immediate Cryotherapy (HPV Test-and-treat) | Arm B: Cytology-based Strategy
Number analyzed (Participants) | 122 | 111
Participants
  Week 26: With hr-HPV Detected | 74 | 78
  Week 52: With hr-HPV Detected: number analyzed (Participants) | 0 | 0
  Week 78: With hr-HPV Detected: number analyzed (Participants) | 0 | 0
  Week 104: With hr-HPV Detected: number analyzed (Participants) | 0 | 0
  Week 130: With hr-HPV Detected: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Arm A: Immediate Cryotherapy (HPV Test-and-treat) vs Arm B: Cytology-based Strategy; Null Hypothesis: There is no difference between Arm A and Arm B with respect to the proportion of participants with hr-HPV at week 26; Test type: Other; p = 0.132, Fisher Exact — [p-value comment as in outcome 5, analysis 1]

7. Secondary Outcome: Number of Participants With High Risk (hr)-HPV by the Xpert HPV Assay at Study Visits.
Description: Number of participants with hr-HPV (HPV 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, 68) as detected by the Xpert HPV assay. Specimens for weeks 52, 78, 104 and 130 were not tested due to insufficient funding.
Time Frame: Weeks 26, 52, 78, 104 and 130 post randomization
Population: Includes participants with results for Xpert HPV assay
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Immediate Cryotherapy (HPV Test-and-treat) | Arm B: Cytology-based Strategy
Number analyzed (Participants) | 119 | 109
Participants
  Week 26: With hr-HPV Detected | 64 | 68
  Week 52: With hr-HPV Detected: number analyzed (Participants) | 0 | 0
  Week 78: With hr-HPV Detected: number analyzed (Participants) | 0 | 0
  Week 104: With hr-HPV Detected: number analyzed (Participants) | 0 | 0
  Week 130: With hr-HPV Detected: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Arm A: Immediate Cryotherapy (HPV Test-and-treat) vs Arm B: Cytology-based Strategy; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.227, Fisher Exact — [p-value comment as in outcome 5, analysis 1]

8. Secondary Outcome: Number of Participants With High Risk (hr)-HPV by the Roche Linear Array HPV Genotyping Test at Study Visits.
Description: Number of participants with hr-HPV (HPV 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, 68) as detected by the Roche Linear Array HPV Genotyping test. Specimens for weeks 52, 78, 104 and 130 were not tested due to insufficient funding.
Time Frame: Weeks 26, 52, 78, 104 and 130 post randomization
Population: Includes participants with results for the Roche Linear Array HPV Genotyping test.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Immediate Cryotherapy (HPV Test-and-treat) | Arm B: Cytology-based Strategy
Number analyzed (Participants) | 92 | 91
Participants
  Week 26: With hr-HPV Detected | 74 | 73
  Week 52: With hr-HPV Detected: number analyzed (Participants) | 0 | 0
  Week 78: With hr-HPV Detected: number analyzed (Participants) | 0 | 0
  Week 104: With hr-HPV Detected: number analyzed (Participants) | 0 | 0
  Week 130: With hr-HPV Detected: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Arm A: Immediate Cryotherapy (HPV Test-and-treat) vs Arm B: Cytology-based Strategy; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 1.000, Fisher Exact — [p-value comment as in outcome 5, analysis 1]

9. Secondary Outcome: Percentage of Participants With Targeted Adverse Events (AEs) Reported Post Cryotherapy in Arm A.
Description: Cryotherapy was performed in Arm A within 7 days of study entry. Targeted AEs four weeks after cryotherapy is provided in the data table below. The AE categories are not mutually exclusive. A participant may have experienced AEs and may be counted in more than one category.
Time Frame: 4 weeks post cryotherapy
Population: Included Arm A participants who had cryotherapy.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Immediate Cryotherapy (HPV Test-and-treat)
Number analyzed (Participants) | 142
percentage of participants
  Profuse watery vaginal discharge | 20
  Mild cervical bleeding | 15
  Heavy odorous discharge | 13
  Cervical infection | 5
  Mild watery vaginal discharge | 4
  Lower Abdominal Pain | 3
  Severe cramps or abdominal pain requiring parenter | 3
  Moderate Watery Vaginal Discharge | 2
  Pelvic inflammatory disease | 1
  Abdominal Pain, Mild, No Medicine Taken | 1
  Had Intermittent Blood Spotting Per Vagina | 1
  Heavy cervical bleeding | 1
  Light Watery Vaginal Discharge | 1
  Mild Odour | 1
  Mild P.V. Spotting | 1
  Mild Vaginal Bleeding | 1
  Mild Vaginal Bleeding Moderate Watery Vaginal Disc | 1
  Minimal Watery Discharge | 1
  Mod Watery Non Offensive Vag Discharge & Mod Yello | 1
  Moderate Offensive Vaginal Watery Discharge | 1
  Moderate Vaginal Discharge | 1
  Moderate Vaginal Watery Discharge And Minimal Yell | 1
  Moderate Vaginal Discharge & Minimal Yellowi | 1
  Post Coital Bleeding | 1
  Moderate Vaginal Watery & Brown Smelly Discharge | 1
  Slight Pv Discharge | 1
  Trichomonas Vaginitis | 1

10. Secondary Outcome: Percentage of Participants With Targeted AEs Reported Post LEEP.
Description: LEEP was performed on participants who had CIN2+. For Arm A participants, LEEP was available starting at week 26; for Arms B and C, LEEP was available starting at study entry. Targeted AEs four weeks after LEEP is provided in the data table below. The AE categories are not mutually exclusive. A participant may have experienced AEs and may be counted in more than one category.
Time Frame: 4 weeks post LEEP
Population: Participants in each arm who had LEEP were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Immediate Cryotherapy (HPV Test-and-treat) | Arm B: Cytology-based Strategy | Arm C : Ineligible for Randomization to Arm A or B
Number analyzed (Participants) | 24 | 34 | 54
percentage of participants
  Cervical bleeding | 50 | 21 | 22
  Vaginal discharge | 12 | 15 | 31
  Cramps or abdominal pain requiring parenteral meds | 12 | 6 | 13
  Vaginal Bleeding | 4 | 3 | 13
  Cervical infection | 0 | 3 | 2
  Metrorrhagia | 4 | 0 | 0
  Pelvic inflammatory disease | 0 | 3 | 0

ADVERSE EVENTS:
Time Frame: AEs reported from entry visit to off study visit (at week 130 or earlier).
Description: At entry, all signs/symptoms (s/s) and lab values Grade >=3 that occurred within 45 days prior to entry were recorded; post entry, s/s and lab values Grade >=3 were recorded. Post entry, all grades of s/s related to cervical cryotherapy or LEEP treatments included in Addendum 1 were reported. SUSAR Reporting Category in DAIDS EAE Manual V2.0 was used. Grading was based on DAIDS AE Grading Table (V1.0) and Addendum 1.
Groups:
- Arm C: Ineligible for Randomization to Arm A or B: Participants were eligible for Arm C under the conditions noted in the inclusion criteria. Participants in Arm C had colposcopy and directed biopsies at entry. If CIN2+ is found by biopsy, then LEEP was performed and a follow-up visit 26 weeks after these procedures was scheduled for the collection of cervical specimens, cytology, and as needed, cervical colposcopy, directed biopsies, and LEEP. After the week 26 visit, Arm C participants went off study.
  Loop Electrosurgical Excision Procedure (LEEP): Participants found to have CIN2+ by biopsy at any point during the study had LEEP, an electro-surgical procedure used to treat high-grade cervical dysplasia.
Arm/Group | Arm A: Immediate Cryotherapy (HPV Test-and-treat) | Arm B: Cytology-based Strategy | Arm C: Ineligible for Randomization to Arm A or B
All-Cause Mortality (participants affected / at risk) | 2/145 | 1/143 | 0/177
Serious Adverse Events (participants affected / at risk) | 5/145 | 2/143 | 5/177
Other Adverse Events (participants affected / at risk) | 60/145 | 49/143 | 38/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Immediate Cryotherapy (HPV Test-and-treat) (N=145) | Arm B: Cytology-based Strategy (N=143) | Arm C: Ineligible for Randomization to Arm A or B (N=177)
Localised infection (Infections and infestations) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Immediate Cryotherapy (HPV Test-and-treat) (N=145) | Arm B: Cytology-based Strategy (N=143) | Arm C: Ineligible for Randomization to Arm A or B (N=177)
Abdominal pain lower (Gastrointestinal disorders) | 14 | 3 | 3
Bacterial vaginosis (Infections and infestations) | 25 | 27 | 9
Cervicitis (Infections and infestations) | 29 | 20 | 27
Cervicitis trichomonal (Infections and infestations) | 9 | 5 | 2
Vulvovaginal candidiasis (Infections and infestations) | 9 | 10 | 3
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 9 | 8 | 3
Cervical dysplasia (Reproductive system and breast disorders) | 12 | 13 | 18
Vaginal discharge (Reproductive system and breast disorders) | 39 | 15 | 15
Vaginal haemorrhage (Reproductive system and breast disorders) | 10 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT01315353/SAP_000.pdf
  • Study Protocol (2015-06-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT01315353/Prot_001.pdf